CLINICAL TRIAL: NCT06348589
Title: Orthostatic Hypotension and Blood Pressure Variability in Persons Undergoing Hemodialysis - an Observational Study
Brief Title: Orthostatic Hypotension and Blood Pressure Variability in Persons Undergoing Hemodialysis
Status: Completed | Type: Observational
Sponsor: Vrinnevi Hospital (Other)
Responsible Party: Principal Investigator, Magnus Wijkman, Principal Investigator, Medically Responsible Physician at the Section for Endocrinology and Diabetology, Vrinnevi Hospital
Other Study IDs: 2023-05959-01
Record Dates: First submitted 2024-03-24; First posted 2024-04-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
High blood pressure is a risk factor for end-stage renal disease and is common in patients undergoing maintenance hemodialysis. Intradialytic hypotension is associated with an adverse prognosis. More knowledge is needed to identify patients at high risk for intradialytic hypotension and dialysis-associated hypotensive episodes. The aim of this observational single-center pilot study is to evaluate whether point-of-care ultrasound measurements may predict intradialytic hypotension and orthostatic blood pressure falls, in patients with chronic kidney disease who undergo maintenance hemodialysis.

DETAILED DESCRIPTION:
Background: Hypertension is an independent risk factor for development of end-stage renal disease and is the leading risk factor for cardiorenal death. It is estimated that more than 80% of patients with end-stage renal disease who undergo maintenance hemodialysis have hypertension. Intensified blood pressure control has been associated with reduced risk of death in patients with hypertension and chronic kidney disease but may increase the risk for intra-dialytic blood pressure falls in patients who undergo hemodialysis. Hemodialysis-associated hypotension has been associated with increased risks for cardiovascular disease and mortality.

Aim: The aim of this observational pilot study is to evaluate whether point-of-care ultrasound measurements may predict intradialytic hypotension and orthostatic blood pressure falls, in patients with chronic kidney disease who undergo maintenance hemodialysis.

Ethics: The study has been approved by the Swedish Ethical Review Authority (2023-05959-01).

Study participants: All patients (n=70) with chronic kidney disease who undergo maintenance hemodialysis at Vrinnevi Hospital in Norrköping, Sweden, will be invited to voluntarily participate in the study. Information about the study will be given orally and in written form. Those who opt to participate will be asked to sign a written informed consent.

Background data collection: For descriptive purposes, information will be collected regarding current and prior medical diagnoses, current medical treatment, anthropometric data, and self-perceived quality of lite (using the validated questionnaire KDQOL-SF). Blood samples will be tested for routine hematological variables, as well as for sodium, potassium, calcium, creatinine, urea and HbA1c.

Ultra-sound measurements: Before initiation of dialysis, point-of-care ultrasound measurements will be performed with the patient resting in a supine position at a 30 degrees angle, using a Sonosite SII ultrasound machine with a curvilinear probe. Measurements of the diameter of the inferior vena cava will be performed at a level approximately 2 cm from the right atrium, and breathing variability of its diameter will be assessed.

Blood pressure measurements: Systolic and diastolic blood pressure measurements will be performed after the patient has been resting for 5 minutes in the supine position, with a cuff size that is appropriate for each patient, with the arm resting at heart level, in the arm where the patient does not have a dialysis fistula, using an automated blood pressure measurement device (Fresenius 6008 CARE System) which is connected to the dialysis equipment. Two measurements (with one minute apart) will be performed 30 minutes before the dialysis session begins, three measurements will be performed after half of the planned dialysis session, and two measurements will be performed 15 minutes after the dialysis session has ended. An orthostatic test, which includes systolic and diastolic blood pressure measurements taken immediately after standing up and 1 and 3 minutes after standing up, will also be performed 30 minutes before the dialysis session begins and 15 minutes after the dialysis session has ended.

Statistics: Background information (demographics, anthropometrics, medical history, medication, biochemical evaluation) will be presented for the entire study population as means with standard deviations, medians with inter-quartile ranges, or as counts with percentages, as appropriate. These variables will also be presented in patients with and without intradialytic blood pressure falls (defined as an intradialytic reduction of systolic blood pressure ≥ 20 mmHg or of diastolic blood pressure ≥10 mmHg), and in patients with and without orthostatic blood pressure falls (defined as an orthostatic reduction of systolic blood pressure ≥ 20 mmHg or of diastolic blood pressure ≥10 mmHg), respectively. Between-group differences will be tested for statistical significance using Student´s t-test, Mann-Whitney U-test, Chi-square test or Fisher´s exact test, as appropriate.

Temporal changes in supine systolic and diastolic blood pressures (assessed prior to dialysis, during dialysis and after dialysis) will be visualized with regression slopes, and mixed models will be used to assess their associations with ultrasound measurements of the inferior vena cava. Associations between ultrasound measurements of the inferior vena cava and the blood pressure changes during the orthostatic blood pressure tests will be visualized with scatter plots and tested for statistical significance with correlation analysis.

The predictive ability of ultrasound measurements of the inferior vena cava and the occurrence of intra-dialytic blood pressure falls and of orthostatic blood pressure falls, respectively, will be assessed with logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing hemodialysis treatment at Vrinnevi Hospital, Norrköping Sweden
* Provision of written informed consent
* Ability to understand instructions and to participate in the investigations

Exclusion Criteria:

* Ongoing acute illness
* Hospitalization within 4 weeks prior to enrollment
* Unability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (n=70) with chronic kidney disease who undergo maintenance hemodialysis at Vrinnevi Hospital in Norrköping, Sweden, will be invited to voluntarily participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Intra-dialytic systolic blood pressure fall of 20 mmHg or larger | Up to 1 week
  Difference between pre-dialytic and intra-dialytic systolic blood pressure
Post-dialytic orthostatic systolic blood pressure fall of 20 mmHg or larger | Up to 1 week
  Change between supine and upright systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Magnus O Wijkman, MD, PhD, Principal Investigator — Vrinnevi Hospital, Department of Internal Medicine, Section of Endocrinology and Diabetology
Locations (1):
- Vrinnevi Hospital, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No